CLINICAL TRIAL: NCT04962997
Title: Health Status of Transgender Women in French Guiana and Paris: a Cross-sectional View (TransGuyane)
Brief Title: Health Status of Transgender Women in French Guiana and Paris (TransGuyane)
Acronym: TransGuyane
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Collaborators: Bichat Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TransGuyane
Record Dates: First submitted 2021-06-09; First posted 2021-07-15 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2021-06

CONDITIONS: Sexual Health; Mental Health
Keywords: Transgender women; Retention in care; Global health; French Guiana
MeSH Terms: conditions — Psychological Well-Being | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transgender women: Major person identifying as a transgender women consulting at Cayenne Hospital (French Guiana) or Bichat Hospital (Paris) between 06/2021 and 10/2022
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Investigator will ensure the completion of a hetero-administered questionnaire which will be carried out in French, English, Portuguese or Spanish depending on the language spoken by the participant, including informations related to Demography and socio-economic conditions, Addictions, Work and studies, Housing, Health coverage, Gender and sexuality, Vulnerabilities and violence, Recourse to care, State of physical health, Mental Health, Prevention and Sexually Transmitted Infections (STIs), Checkup, Transition path and clinical complications and Dermatological problems.
  Investigator will collect the data relating to the clinical examination, dermatological examination and the search for STIs (blood and / or urine) carried out in the routine care of the participant in a case report form (CRF).
  The estimated duration of the interviews and the consultation is approximately 1 hour and 30 minutes per patient.

SUMMARY:
Assessing and comparing the life and health status of transgender or trans women in French Guiana and Paris. Conducting a questionnaire on physical, mental and sexual health, migration history, transition, and STI screening.

DETAILED DESCRIPTION:
Transgender or trans women in French Guiana are not known to the hospital environment and rarely seek care: only about fifteen patients are followed up in the Infectious and Tropical Diseases Unit (UMIT) and the Adult Day Hospital (HDJA) of the Cayenne Hospital Center for Human Immunodeficiency Virus (HIV) infection. There is therefore a lack of knowledge of this population, of their health needs (physical, sexual and mental) but also a lack of assistance in the transition process. However, the violence suffered and the risks of infection are high among transgender women who frequently resort to sex work. In fact, they are said to carry the highest burden of HIV in the world, particularly in South America. The need for HIV prevention among transgender women in South America is great.

There is no bibliography of published works concerning transgender women in French Guiana, whereas there are more and more publications from countries that are geographically close (Brazil, Peru, United States), or even from metropolitan France. It is therefore necessary to address this issue in French Guiana. The population of transgender women followed up at the Bichat Hospital (for HIV infection or as part of a sexual health follow-up) represents one of the largest active files of transgender women in France and offers the opportunity to look at these two populations from a cross-sectional perspective.

The study will be cross-sectional and multicentric (Cayenne in French Guiana, Paris) and will include transgender women who have reached the age of majority and who agree to answer a questionnaire concerning their living and socio-economic conditions, their migration, their physical, sexual and mental health, and their transition process. Data relating to the search for Sexually Transmitted Infection STIs check-up as well as dermatological examination will be studied in particular with the agreement of the participants.

Data relating to the second consultation will be studied in particular (report of results) without systematic follow-up.

Non-interventional research (RIPH category 3). Cross-sectional observational multicentric study: at the CHC (Cayenne, French Guiana) and at Bichat Hospital (Paris).

ELIGIBILITY:
Inclusion Criteria:

* Person identifying as a transgender woman
* Consulting at Cayenne Hospital (French Guiana) or Bichat Hospital (Paris)
* Between 07/2021 and 10/2022
* Major
* No opposition to the study
* Absence of neurological or psychiatric disorders that prevented understanding of the study and free participation (sequelae of cerebral toxoplasmosis with aphasia, deaf and mute person, active neuro-meningeal opportunistic infections with cognitive impairment…)

Exclusion Criteria:

* Minor
* Refusal to participate and/or neurological or psychiatric disorder preventing understanding of the study
* Not be able to answer questions in languages mastered by principal investigator (French, English, Spanish or Portuguese)
* Person under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender women
Study Population: Person identifying as a transgender woman consulting at Cayenne Hospital (French Guiana) or Bichat Hospital (Paris) between 07/2021 and 10/2022
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Describe the frequency of violence suffered by transgender women treated in Cayenne or Paris | Day 0
  Frequency of psychological, physical and sexual violence suffered by transgender women

SECONDARY OUTCOMES:
Describe the state of health of transgender women in Cayenne and Paris | Day 0
  Describe the state of health of transgender women based on the data collected
Compare these results with those of the National Survey of Transgender Women Living with Human Immunodeficiency Virus | 17 months
  Compare these results with those of the National Survey of Transgender Women Living with Human Immunodeficiency Virus (Dr. Spire's Metropolitan Study on "Trans identity and Human Immunodeficiency Virus").
Describe the state of health of transgender women in Cayenne and Paris | Day 1
  Describe the state of health of transgender women based on the data collected

CONTACTS AND LOCATIONS:
Overall Officials: Chloé BERTIN, Principal Investigator — Centre Hospitalier de Cayenne
Locations (2):
- Centre Hopsitalier Uiversitaire de Bichat, Paris, France
- Centre Hospitalier de Cayenne, Cayenne, Guyane Française, French Guiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baral SD, Poteat T, Stromdahl S, Wirtz AL, Guadamuz TE, Beyrer C. Worldwide burden of HIV in transgender women: a systematic review and meta-analysis. Lancet Infect Dis. 2013 Mar;13(3):214-22. doi: 10.1016/S1473-3099(12)70315-8. Epub 2012 Dec 21. PMID 23260128
- [Background] Grinsztejn B, Jalil EM, Monteiro L, Velasque L, Moreira RI, Garcia AC, Castro CV, Kruger A, Luz PM, Liu AY, McFarland W, Buchbinder S, Veloso VG, Wilson EC; Transcender Study Team. Unveiling of HIV dynamics among transgender women: a respondent-driven sampling study in Rio de Janeiro, Brazil. Lancet HIV. 2017 Apr;4(4):e169-e176. doi: 10.1016/S2352-3018(17)30015-2. Epub 2017 Feb 8. PMID 28188030
- [Background] Silva-Santisteban A, Eng S, de la Iglesia G, Falistocco C, Mazin R. HIV prevention among transgender women in Latin America: implementation, gaps and challenges. J Int AIDS Soc. 2016 Jul 17;19(3 Suppl 2):20799. doi: 10.7448/IAS.19.3.20799. eCollection 2016. PMID 27431470
- [Background] Baggaley RF, White RG, Boily MC. HIV transmission risk through anal intercourse: systematic review, meta-analysis and implications for HIV prevention. Int J Epidemiol. 2010 Aug;39(4):1048-63. doi: 10.1093/ije/dyq057. Epub 2010 Apr 20. PMID 20406794
- [Background] Operario D, Burton J, Underhill K, Sevelius J. Men who have sex with transgender women: challenges to category-based HIV prevention. AIDS Behav. 2008 Jan;12(1):18-26. doi: 10.1007/s10461-007-9303-y. Epub 2007 Aug 19. PMID 17705095
- [Background] Pinto RM, Melendez RM, Spector AY. Male-to-Female Transgender Individuals Building Social Support and Capital From Within a Gender-Focused Network. J Gay Lesbian Soc Serv. 2008 Sep 1;20(3):203-220. doi: 10.1080/10538720802235179. PMID 20418965
- [Background] Reisner SL, Poteat T, Keatley J, Cabral M, Mothopeng T, Dunham E, Holland CE, Max R, Baral SD. Global health burden and needs of transgender populations: a review. Lancet. 2016 Jul 23;388(10042):412-436. doi: 10.1016/S0140-6736(16)00684-X. Epub 2016 Jun 17. PMID 27323919
- [Background] Poteat T, Wirtz AL, Radix A, Borquez A, Silva-Santisteban A, Deutsch MB, Khan SI, Winter S, Operario D. HIV risk and preventive interventions in transgender women sex workers. Lancet. 2015 Jan 17;385(9964):274-86. doi: 10.1016/S0140-6736(14)60833-3. Epub 2014 Jul 22. PMID 25059941
- [Background] Operario D, Soma T, Underhill K. Sex work and HIV status among transgender women: systematic review and meta-analysis. J Acquir Immune Defic Syndr. 2008 May 1;48(1):97-103. doi: 10.1097/QAI.0b013e31816e3971. PMID 18344875
- [Background] Ferreira S Jr, Francisco PMSB, Nogueira PA. [Profile of transvestites and transgender women: tuberculosis and HIV/AIDS in the city of Sao Paulo]. Rev Panam Salud Publica. 2016 Dec;40(6):410-417. Portuguese. PMID 28718489
- [Background] Zoni AC, Gonzalez MA, Sjogren HW. Syphilis in the most at-risk populations in Latin America and the Caribbean: a systematic review. Int J Infect Dis. 2013 Feb;17(2):e84-92. doi: 10.1016/j.ijid.2012.07.021. Epub 2012 Oct 12. PMID 23063547
- [Background] Solomon MM, Mayer KH, Glidden DV, Liu AY, McMahan VM, Guanira JV, Chariyalertsak S, Fernandez T, Grant RM; iPrEx Study Team. Syphilis predicts HIV incidence among men and transgender women who have sex with men in a preexposure prophylaxis trial. Clin Infect Dis. 2014 Oct;59(7):1020-6. doi: 10.1093/cid/ciu450. Epub 2014 Jun 13. PMID 24928295
- [Background] Keshinro B, Crowell TA, Nowak RG, Adebajo S, Peel S, Gaydos CA, Rodriguez-Hart C, Baral SD, Walsh MJ, Njoku OS, Odeyemi S, Ngo-Ndomb T, Blattner WA, Robb ML, Charurat ME, Ake J; TRUST/RV368 Study Group. High prevalence of HIV, chlamydia and gonorrhoea among men who have sex with men and transgender women attending trusted community centres in Abuja and Lagos, Nigeria. J Int AIDS Soc. 2016 Dec 7;19(1):21270. doi: 10.7448/IAS.19.1.21270. eCollection 2016. PMID 27931519
- [Background] Wickersham JA, Gibson BA, Bazazi AR, Pillai V, Pedersen CJ, Meyer JP, El-Bassel N, Mayer KH, Kamarulzaman A, Altice FL. Prevalence of Human Immunodeficiency Virus and Sexually Transmitted Infections Among Cisgender and Transgender Women Sex Workers in Greater Kuala Lumpur, Malaysia: Results From a Respondent-Driven Sampling Study. Sex Transm Dis. 2017 Nov;44(11):663-670. doi: 10.1097/OLQ.0000000000000662. PMID 28708696
- [Background] Kojima N, Park H, Konda KA, Joseph Davey DL, Bristow CC, Brown B, Leon SR, Vargas SK, Calvo GM, Caceres CF, Klausner JD. The PICASSO Cohort: baseline characteristics of a cohort of men who have sex with men and male-to-female transgender women at high risk for syphilis infection in Lima, Peru. BMC Infect Dis. 2017 Apr 11;17(1):255. doi: 10.1186/s12879-017-2332-x. PMID 28399798